CLINICAL TRIAL: NCT06070363
Title: Effectiveness of Manual Acupuncture and Standard Therapy Compared to Standard Therapy in Gynecological Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Suryamin Suryamin, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-06-1047
Record Dates: First submitted 2023-08-31; First posted 2023-10-06 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Gynecologic Cancer; Cancer Related Pain; Cancer Pain; Acupuncture
Keywords: acupuncture; Manual Acupuncture; Cancer Pain; Cancer Related Pain; Gynecologic Cancer
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator blind the participant allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The Patient are cancer patient that experience cancer pain that only receive analgetic drug treatment according to WHO Stepledder of Pain
- Manual acupuncture and standard Therapy (Experimental): The Patient are cancer patient that experience cancer paint that receive analgetic drug treatement according WHO stepledder of pain and receive manual acupuncture
  Interventions: Other: Manual Acupuncture

INTERVENTIONS:
Other: Manual Acupuncture — Acupuncture Needle Insertion
  Arms: Manual acupuncture and standard Therapy

SUMMARY:
Cancer patients experience cancer pain as much as 66%. Cancer pain is pain that occurs in patients with neoplastic/malignancy and the source of the pain can come from malignant processes, treatments such as radiotherapy, chemotherapy, and surgery as well as other causes that are not related to malignancy processes. Unresolved pain can reduce the quality and life expectancy of cancer pain patients. The prevalence of cancer itself in Indonesia, the case of cervical cancer itself ranks second after breast cancer. In recent decades, acupuncture analgesics have been widely used to relieve cancer pain, and can also reduce the dose and side effects of analgesics. However, substantially the use of acupuncture in cancer pain is still very rare.

DETAILED DESCRIPTION:
The main outcome is to analyze the effectiveness of manual acupuncture therapy (LI4,PC6, LR3,ST36, and SP6 plus standard therapy on pain intensity (VAS score), changes in analgesic dose, and quality of life (QLQ C-30 EORTC score) in patients with gynecological cancer pain compared to standard therapy alone.

The patient will attempt 3-day manual acupuncture therapy with seven days follow up Patient will receive acupuncture therapy daily for 3 days, for 15 minute each day.

The research design in this study was a single-blinded randomized control clinical trial. With outcome measures for

With Subject criteria:

Inclusion Criteria

1. The patient is diagnosed with gynecological cancer
2. Women over 18 years to 65 years
3. Subjects experiencing cancer pain, with VAS ≥4, namely pain caused by:

   * tumors,
   * before or during a therapeutic process (radiation therapy, chemotherapy, or post-surgery)
   * side effect or the result of toxicity of cancer treatment
   * Supportive therapy (palliative therapy, painkillers, antidepressants)
4. Willing to participate in this study and sign an informed consent Exclusion Criteria

1) The patient has a medical emergency / hemodynamically unstable 2) Patients with contraindications for manual acupuncture procedures such as wounds and infections at the point where the puncture will be performed, patients allergic to stainless steel62 3) Uncooperative patients (patients with negative and aggressive affect, who do not allow acupuncture therapy) 4) There is a tumor in the area that will be stabbed and stimulated in the pregnant woman's abdomen, close to the heart, or around the carotid sinus, lymphedema, needle insertion into the prosthesis 5) Patients with heart rhythm disorders 6) The patient uses a pacemaker 7) Patients with disorders of the auricle such as eczema, external otitis, and psoriasis 8) Patients with blood clotting disorders, with platelets <50,000, and in neutropenic conditions with neutrophils <1000

ELIGIBILITY:
Inclusion Criteria:

* Female 18 to 65 years old
* Gynecocal cancer with pain ≥ 4 acording Visual Analog scale and receive analgetic medicine
* The pain cause by

  1. direct from cancer
  2. Treatment proces surgery, radiotherapy, chemotherapy, paliatif treatment, supportive treatment
  3. Adverse reaction form treatment and intoxication

Exclusion Criteria:

* emergency case patient with hemodynamic instable
* patient with uncooperative behavior because ith serious psychological disorders, no currently undergoing psychiatric treatment, aggressive behavior, that not allowed for acupuncture.
* Patients with blood clotting disorders, with platelets <50.000 and in neutropenic condition with <1000 neutrophils.

The patient has an allergy to stainless steel acupuncture needles. Wounds at the acupuncture point puncture sites, skin infections in the ears. On patients with eczema on the ears, external otitis or psoriasis.

There is a tumor in the area that will be stabbed and stimulated in the stomach pregnant women, close to the heart, or in the area of the carotid sinus lymphedema, insertion into the prosthesis.

Patients with heart rhythm disorders. The patient uses a pace maker.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with gynecology cancer
Enrollment: 58 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Pain severity with Visual Analog Scale | Before treatment, After treatment in day 1, day 2, day 3, day 5 and day 7
  Visual Analog Scale (VAS) that score 0 is no pain to 100 the worse pain A higher scale means worse outcomes

SECONDARY OUTCOMES:
Quality of Life with European Organisation for Research and Treatment of Cancer Quality of Life C30 | before treatment and 7 day after treatment
  European Organisation for Research and Treatment of Cancer Quality of Life C30, that include two item of review functional scale and the global health scale both scale the higher the score the outcome will be better
Analgetic Usage in dosage and frequency | Before treatment, After treatment in day 1, day 2, day 3, day 5 and day 7
  Description of analagetic dosage and frequency during observation that will be describe as medicine category opioid non opioid, dosage and frequency

CONTACTS AND LOCATIONS:
Overall Officials: Suryamin Suryamin, Study Director — Indonesia University
Locations (4):
- Indonesia (4):
  - Fatmawati Hospital, Jakarta, Dki Jakarta
  - Persahabatan Hospital, Jakarta, Dki Jakarta
  - Suryamin Hung, Jakarta, DKI Jakarta
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, Dki Jakarta

IPD SHARING:
Plan to Share IPD: No